CLINICAL TRIAL: NCT03724045
Title: Back Side of the Moon Study: What is the Efficiency of Nutritional Therapy (Calories and Nitrogen) in ICU and on the Ward and What is the Metabolic Profile of Patients After ICU? Could Supplemental Nutrition Fill the Gap?
Brief Title: Back Side of the Moon: Nutritional Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Elisabeth De Waele, Prof. Dr., Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BUN 143201837553
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Nutritional Deficiency; Hospitalism
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Back Side of the Moon (Experimental): Patients will be screened and enrolled at the ICU. Extraordinary measurements concerning nutritional status will be performed, to investigate whether patients at the ICU actually meet their nutritional needs. The same patients as above will be followed up, once discharge from ICU to a low-care ward has taken place. From there, they will be followed up until discharge from the hospital. The procedures are the same as in the ICU. The results obtained at the low-care ward will be compared to those from the ICU. 6 months after hospital discharge, morbidity and mortality will be assessed.
  A substudy of included COVID-19 positive patients will be analysed and compared to non COVID-19 patients.
  Interventions: Dietary Supplement: Back Side of the Moon

INTERVENTIONS:
Dietary Supplement: Back Side of the Moon — The procedures are: several measurements will be performed, including some which are not part of the Standard Operating Procedure, hence causing it to be considered interventional.
  Follow-up during consultation on pneumology until max. 6 months post-admission on the ICU.

SUMMARY:
Prospective observational follow-up of Intensive Care Unit (ICU) survivors on the adequacy of nutritional therapy: what is the mean caloric and nitrogen intake and how does their metabolic profile evolve over time? Is supplemental nutrition, in any forms, indicated to fill the caloric and protein gap? Would IV access be a barrier for SPN, and would subcutaneous parenteral nutrition be welcomed by health care practitioners and patients? Are patient centered outcomes (physical function, quality of life, performance in activities of daily living) correlated with nutritional adequacy and metabolic profile? Overall: are ICU survivors well fed after they leave ICU until hospital discharge? What kind of nutrition would possibly be useful to optimize the intake? How do their energy and protein requirements evolve? What is the physical and mental status of ICU survivors and is this correlated with nutritional status?

DETAILED DESCRIPTION:
Nutritional therapy has been a matter of debate for several decades. Patient selection, time point of intervention, dosing of calories, protein, vitamins and trace elements and route of artificial nutrition have been the subject of research initiatives, and although consensus exist on several matters, some questions remain unanswered.

At the same time length of ICU stay is shortening, and ICU survivors know an extended hospital stay in the ward. The window of opportunity for adequate nutritional therapy is thereby divided between the critically ill department and the ward. Little is known on the metabolic evolution of ICU survivors, and some data support an increased protein and calorie need post resuscitation to attenuate lean body mass and promote recovery. Adequate protein and calorie delivery is required to facilitate recovery. Nevertheless, adherence to nutrition guidelines seems to be difficult in the resource-dens environment of ICU, as proven by data from the 'Nutritionday' project. Adequacy of nutritional therapy management for ICU patients that are discharged to the ward is unknown. Fair nutritional therapy could be discovered by this trial, but the possibility exists that crude iatrogenic malnutrition is discovered. This information would act as baseline data to build nutritional quality improvement programs, using different forms of artificial nutrition, from oral supplements over enteral and parenteral nutrition.

Secondly, metabolic information on ICU survivors is scarce. Body weight is often poorly followed-up, body composition evolution, including phase angle, is unknown, and metabolic monitoring by indirect calorimetry could reveal changed metabolic state and substrate use defined by the respiratory quotient.

Thirdly, relevant barriers to the use of an intravenous access have been reported: patients who are agitated or confused or where the placement and/or maintenance of an (central) IV line would cause suffering or pain. These patients show to be low in numbers, but nutrition could possibly be restrained . This raises an interesting question on the access issue. The enteral route has to be focused on, as information on patients' experience is available in home enteral nutrition, but data in post critical illness patients is non-existing. Clinical practices in the field of nutrition can be influenced by behavioral patterns of health care practitioners and patients. A questionnaire will be used to evaluate opinions of health care practitioners and patients. This information could be of value for the way we look at nutritional management.

This project targets the evaluation of nutritional adequacy on ICU and in the ward, and the observation of metabolic evolution of ICU survivors. Nutritional adequacy and metabolic profile will be investigated in correlation to patient centered outcomes (physical function, quality of life, performance in activities of daily living).

A substudy of included COVID-19 positive patients will be analysed and compared to non COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 7 days ICU stay
* ≥ 7 days hospital stay

Exclusion Criteria:

* < 7 days ICU stay
* metabolic disease
* restriction on nutritional therapy due to comorbid disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Morbidity | 6 months after hospital discharge
  Morbidity

SECONDARY OUTCOMES:
Mortality | 6 months after hospital discharge
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth De Waele, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No
Described in the study contract by the main sponsor:
  Upon completion of the Study, the INSTITUTION and INVESTIGATOR will seek to publish the results of the Study in a peer-reviewed literature. BAXTER Confidential Information shall not be disclosed without prior written permission from BAXTER. For purposes of this Agreement, "Publication" shall mean any paper, article, manuscript, report, poster, internet posting, presentation slides, abstract outline, video, instructional material, presentation (in the form of a written summary), or other public disclosure of the results of the Study, in printed, electronic, oral or other form.

REFERENCES:
- [Background] Preiser JC, van Zanten AR, Berger MM, Biolo G, Casaer MP, Doig GS, Griffiths RD, Heyland DK, Hiesmayr M, Iapichino G, Laviano A, Pichard C, Singer P, Van den Berghe G, Wernerman J, Wischmeyer P, Vincent JL. Metabolic and nutritional support of critically ill patients: consensus and controversies. Crit Care. 2015 Jan 29;19(1):35. doi: 10.1186/s13054-015-0737-8. PMID 25886997
- [Background] Wischmeyer PE. Tailoring nutrition therapy to illness and recovery. Crit Care. 2017 Dec 28;21(Suppl 3):316. doi: 10.1186/s13054-017-1906-8. PMID 29297385
- [Background] Bendavid I, Singer P, Theilla M, Themessl-Huber M, Sulz I, Mouhieddine M, Schuh C, Mora B, Hiesmayr M. NutritionDay ICU: A 7 year worldwide prevalence study of nutrition practice in intensive care. Clin Nutr. 2017 Aug;36(4):1122-1129. doi: 10.1016/j.clnu.2016.07.012. Epub 2016 Aug 9. PMID 27637833
- [Background] Caccialanza R, Constans T, Cotogni P, Zaloga GP, Pontes-Arruda A. Subcutaneous Infusion of Fluids for Hydration or Nutrition: A Review. JPEN J Parenter Enteral Nutr. 2018 Feb;42(2):296-307. doi: 10.1177/0148607116676593. Epub 2017 Dec 20. PMID 29443395
- [Background] Lim ML, Yong BYP, Mar MQM, Ang SY, Chan MM, Lam M, Chong NCJ, Lopez V. Caring for patients on home enteral nutrition: Reported complications by home carers and perspectives of community nurses. J Clin Nurs. 2018 Jul;27(13-14):2825-2835. doi: 10.1111/jocn.14347. Epub 2018 Apr 22. PMID 29518266